CLINICAL TRIAL: NCT03408301
Title: The Effects of Sympathovagal Balance Before Tourniquet Deflation on a Decrease in Arterial Blood Pressure Following the Deflation During Total Knee Replacement Arthroplasty
Brief Title: The Status of Autonomic Tone Before Tourniquet Deflation During Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, JongHae Kim, Associate Professor, Daegu Catholic University Medical Center
Other Study IDs: CR-13-071
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Hypotension; Blood Pressure, Low
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tourniquet deflation: Tourniquet deflation after insertion of the prosthetic components during total knee replacement arthroplasty under spinal anesthesia
  Interventions: Procedure: Tourniquet deflation

INTERVENTIONS:
Procedure: Tourniquet deflation — Tourniquet deflation

SUMMARY:
This study evaluates the influences of the status of sympathovagal balance before tourniquet deflation on a decrease in arterial blood pressure following the deflation during total knee replacement arthroplasty

DETAILED DESCRIPTION:
Patients present with different hemodynamic profiles after intraoperative tourniquet deflation during total knee replacement arthroplasty.

Sympathovagal balance can be measured before tourniquet deflation and might determine the hemodynamic response to tourniquet deflation.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists physical status I - II
2. Body mass index < 35 kg/m2

Exclusion Criteria:

1. Coagulation deficiencies
2. Known allergies to local anesthetics
3. Neurologic deficit on the side being operated on
4. Inflammation at the lumbar puncture site
5. Cardiac conduction disorders or arrhythmias
6. Congestive heart failure
7. Serum electrolyte abnormalities
8. Psychiatric disorders
9. Patient's refusal
10. Difficulty communicating with medical personnel
11. Severe hypovolemia
12. Increased intracranial pressure
13. Severe aortic stenosis
14. Severe mitral stenosis

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total knee replacement arthroplasty in a tertiary university hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2014-07-29 (Actual); Study Completion 2014-07-30 (Actual)

PRIMARY OUTCOMES:
Sympathovagal balance | During 5 minutes before tourniquet deflation
  The ratio of low-to-high frequency power of heart rate variability calculated from the 5-minute long electrocardiogram waveform

SECONDARY OUTCOMES:
Noninvasive hemodynamic parameters | During 5 minutes before tourniquet deflation
  Average cardiac index
Maximum percent change in mean arterial blood pressure | During 10 minutes after tourniquet deflation
  The discrepancy between minimum mean arterial blood pressure after tourniquet deflation and mean arterial blood pressure immediately before tourniquet deflation, which is divided by mean arterial pressure immediately before tourniquet deflation

CONTACTS AND LOCATIONS:
Overall Officials: JongHae Kim, M.D., Principal Investigator — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No